CLINICAL TRIAL: NCT04891211
Title: Evaluation of Retinal Structure in Pediatric Subjects With Vitamin D Deficiency
Brief Title: Retinal Changes in Vitamin D Deficiency
Acronym: VDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, Emre Aydemir, Principal Investigator, Adiyaman University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: EA180919
Record Dates: First submitted 2021-05-11; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Pediatric Disorder; Vitamin D Deficiency; Retinal Disease; Choroidal Disease; Optic Nerve Diseases
MeSH Terms: conditions — Vitamin D Deficiency; Retinal Diseases; Choroid Diseases; Optic Nerve Diseases

STUDY DESIGN:
Intervention Model Description: Group 1: 1) age <18 years old; 2) serum vitamin D [(25(OH) D), calcitriol] level <20 ngr/mL in previous two weeks Group 2: 1) age <18 years old; 2) serum vitamin D [(25(OH) D), calcitriol] level >20 ngr/mL in previous two weeks
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patients will be examined without knowing their vitamin D level. The OCT evaluations will be performed by a highly trained ophthalmic technician, and the compatibility of the results will be confirmed by two experienced retinal specialists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric endocrinologist (Active Comparator): Patient selection by pediatric endocrinologist on the basis of vitamin D
  Interventions: Dietary Supplement: Vitamin D deficiency
- Ophthalmologist (No Intervention): 1. Evaluation of the results by 2 different retina specialists during the examination of patients
  2. Interpretation of the results without knowing the vitamin D level of patients

INTERVENTIONS:
Dietary Supplement: Vitamin D deficiency — Ocular significance of vitamin D deficiency in pediatric cases
  Arms: Pediatric endocrinologist

SUMMARY:
Retinal tissue parameters of pediatric patients with vitamin D deficiency will be evaluated in this prospective case-control study. The patients will be divided into 2 groups according to the vitamin D level. Retinal vessel diameters, retinal nerve fiber evaluation, choroidal thickness will be evaluated. Choroidal thinning decrease in retinal artery diameter and increase in retinal vein diameter will be detected in the vitamin D deficiency group.

DETAILED DESCRIPTION:
The study of the relationship between vitamin D status and retinal diseases is a new concept, and there is a large gap in research focusing on the pediatric population in the literature. The importance of vitamin D in retinal maturation and its role in the development of retinal diseases at a young age is being investigated. In this sense, as far as known, it is the first study investigating retinal structure parameters in pediatric patients with vitamin D deficiency.

ELIGIBILITY:
Inclusion Criteria:(Group 1):

1. age <18 years old
2. serum vitamin D [(25(OH) D), calcitriol] level <20 ngr/mL in previous two weeks
3. visual acuity >20/20
4. manifest refraction spherical equivalent <3D
5. normal biomicroscopic and fundus examination.

Exclusion Criteria:

1. history of any chronic ocular diseases, except for refractive error (e.g., uveitis, glaucoma, retinopathy of prematurity)
2. history of ocular surgery (e.g., cataract, strabismus, open globe injury, laser photocoagulation)
3. having an ocular abnormality (e.g., persistent fetal vasculature, optic disc hypoplasia, fovea plana)
4. history of systemic diseases that have the potential to affect ocular tissues (e.g., diabetes mellitus, Graves' disease, albinism, Down syndrome, Fabry diseases, Wilson syndrome)
5. history of any systemic diseases that can affect the serum vitamin D level (e.g., parathormone or calcium metabolism disorders)
6. already receiving vitamin D treatment.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Pediatrics population
Enrollment: 150 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
choroidal thickness | up to 3 months
  subfoveal, and subfoveal 1500-µm- and 3000-µm-diameter distance nasal and temporal areas
retinal nerve fiber layer | up to 3 months
  Retinal nerve fiber layer will be detected by optical coherence tomography
The central retinal artery and vein calibers | up to 3 months
  The central retinal artery and vein calibers will be analyzed with the Interactive Vessel Analyzer

SECONDARY OUTCOMES:
blood vitamin D levels | up to 3 months
  vitamin D deficiency or normal effects of vitamin D deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Emre Aydemir, M.D., Principal Investigator — Adiyaman University
Locations (1):
- Adıyaman U, Adıyaman, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Participants will be told what the plan provided and how it worked. Information will be given about when he will participate in the study and the measurements to be taken for the study.
  It will be emphasized that there was nothing that harmed the participants in the examinations.
Supporting Information: Study Protocol, ICF
Time Frame: Participants will be examined at same times of the day in order not to affect the measurement results.
Access Criteria: Participants will be divided into groups according to their vitamin D levels

REFERENCES:
- [Result] Poon M, Craig ME, Kaur H, Cusumano J, Sasongko MB, Wong TY, Donaghue KC. Vitamin D deficiency is not associated with changes in retinal geometric parameters in young people with type 1 diabetes. J Diabetes Res. 2013;2013:280691. doi: 10.1155/2013/280691. Epub 2013 Jul 7. PMID 23936865